CLINICAL TRIAL: NCT03128788
Title: Comparison of Extent of Epidurography and Thoracic Epidural Pressure in the Prone and Lateral Decubitus Position
Brief Title: Comparison of Thoracic Epidural Pressure in the Prone and Lateral Decubitus Position
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, Ji Hee Hong, Professor, Keimyung University Dongsan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-12-048
Record Dates: First submitted 2017-04-20; First posted 2017-04-25 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Thoracic Epidural Injection
Keywords: epidurography epidural pressure patient posture

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Comparator: supine position (Active Comparator): Active Comparator: supine position thoracic epidural catheterization with supine position
  Interventions: Procedure: thoracic epidural catheterization
- Active Comparator: flexed lateral position (Active Comparator): Active Comparator: flexed lateral position thoracic epidural catheterization with flexed lateral position
  Interventions: Procedure: thoracic epidural catheterization

INTERVENTIONS:
Procedure: thoracic epidural catheterization — thoracic epidural catheterization thoracic epidural catheterization for the management of postoperative pain

SUMMARY:
It is reported that the distribution of contrast medium had an obvious correlation with the extent of sensory analgesia after injection of LA. Our previous study showed that different posture (prone vs. lateral decubitus) resulted in different degree of contrast medium spread. We supposed that differences of epidural pressure between diverse postures might be one factor contributing those differences of epidurography.

This study was designed to compare the epidural pressure and extent of spread of epidurography between prone and lateral decubitus position

DETAILED DESCRIPTION:
It is known that postoperative pain after thoracotomy or lobectomy is very severe, therefore, intraoperative or postoperative pain management using continuous thoracic epidural catheterization is suggested good option to prevent this potential complication.

The spread of local anesthetics is influenced by various factors including volume, location of needle insertion, speed of injection, patient position, age, weight and height. However, there are few studies about the effect of different patient position affeting the epidural pressure and the extent of spread of contrast medium during thoracic epidural catheterization.

Studies of lumbar epidural blockade have shown that lateral position can produce 0-3 segment more to the dependent position compared to the supine position. When the same amount of local anesthetic was injected in supine of sitting position, the most cephalad level of spread was indifferent. Recent studies showed that neck flexion demonstrated significant cephalad spread of contrast dye in high thoracic epidural blockade. The purpose of this study was to compare and evaluate the changes of epidural pressure with extent of spread of contrast medium between different posture

ELIGIBILITY:
Inclusion Criteria:

* lung cancer
* liver cancer
* stomach cancer
* pancreas cancer

Exclusion Criteria:

* coagulopathy
* infection
* previous spine fusion at thoracic level

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2018-01-02 (Actual); Study Completion 2018-02-02 (Actual)

PRIMARY OUTCOMES:
Epidural pressure | 15 minutes after the completion of the intervention
  Epidural pressure (mmHg) measurement using pressure transducer between different posture

SECONDARY OUTCOMES:
Contrast dye assessment | 5 minutes after the completion of the intervention
  Number of segment convered by contrast dye assessed through fluoroscopic image

CONTACTS AND LOCATIONS:
Overall Officials: Ji Hee Hong, PhD, Principal Investigator — Keimyung University
Locations (1):
- Ji Hee Hong, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No